CLINICAL TRIAL: NCT00173225
Title: Association Between Sputum and Plasma Levels of Nociceptin and Substance P With Cough Severity and Airway Hyperreactivity in Patients With Asthma, COPD and Chronic Cough
Brief Title: Sputum and Plasma Levels of Nociceptin and Substance P in Patients With Asthma, COPD and Chronic Cough
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700531
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Asthma; COPD; Cough
Keywords: nociceptin; sunstance P; asthma; COPD; cough
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Cough

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The aims of this study are to investigate the association between sputum and plasma levels of nociceptin and substance P with cough severity and airway hyperreactivity in patients with asthma, COPD and chronic cough.

DETAILED DESCRIPTION:
Recent animal studies have found that nociceptin can inhibit cough responses induced by capsaicin. We hypothesize that sputum and plasma levels of these peptides may reflect some neurochemical alterations in airway cough reflex or neurogenic inflammation in asthma or COPD. The aims of this study are to investigate the association between sputum and plasma levels of nociceptin and substance P with cough severity and airway hyperreactivity in patients with asthma, COPD and chronic cough. We will enroll 260 patients (100 patients with asthma, 60 with COPD and 100 with chronic cough) as well as 40 healthy subjects for this study. Sputum and peripheral blood will be collected and concentrations of nociceptin and substance P will be measured by ELISA. These levels will be correlated with cough severity (symptom scores), and airway hyperresponsiveness to inhaled methacholine as measured by PC20. Sputum and plasma concentrations of both peptides will be rechecked after clinical improvements in cough or airway symptoms are achieved after therapy.

ELIGIBILITY:
Inclusion Criteria:patients with asthma, COPD, chronic cough

-

Exclusion Criteria:patients refusing blood sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-06; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hung Kuo, MD, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- Ping-Hung Kuo, Taipei, Taiwan